CLINICAL TRIAL: NCT00751699
Title: A Randomized, Open-label, Multiple Dose, Parallel Group Study to Evaluate 5 ASA and N Ac 5 ASA Pharmacokinetics Following Administration of Oral Doses of Asacol 2.4 g/Day and Lialda 2.4 g/Day for 7 Days in Healthy Volunteers
Brief Title: Pharmacokinetics of Asacol 2.4 g/Day and Lialda 2.4 g/Day in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007011
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Asacol 6x400 mg Q24h at 7 am for 7 days
  Interventions: Drug: Asacol
- 2 (Experimental): Asacol 2x400 mg Q8h at 7 am, 3 pm, and 11 pm for 7 days
  Interventions: Drug: Asacol
- 3 (Experimental): Lialda 2x1.2g Q24h at 7 am for 7 days
  Interventions: Drug: Lialda

INTERVENTIONS:
Drug: Asacol — Asacol tablets, 6 tablets per day at 7 am for 7 days
  Arms: 1
Drug: Asacol — Asacol tablets, 400 mg, 2 tablets at 7 am, 3 pm, and 11 pm for 7 days
  Arms: 2
Drug: Lialda — Lialda tablets 1.2 g, 2 tablets once a day at 7 am for 7 days
  Arms: 3

SUMMARY:
This study evaluated pharmacokinetics of 5-ASA and N-Ac-5-ASA associated with each of 3 regimens of oral mesalamine 2.4 g/day (Lialda 2.4 g/day 2 x 1.2 g every 24 hours, Asacol® 6 x 400 mg every 24 hours, or Asacol 2 x 400 mg every 8 hours). Primary endpoints were 5-ASA area under the plasma concentration versus time curve from zero to 24 hours (AUC24) and total 5-ASA percent of dose excreted (A'e [%]) over the 24-hour period on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years of age, inclusive, at screening and in good general health based on medical history, physical examination, and laboratory evaluation;
* If female, must be (as documented by patient reported medical history):
* postmenopausal (at least 1 year without spontaneous menses), or
* surgically sterile (tubal ligation or hysterectomy), or
* using acceptable contraception [e.g., sexual partner with non-reversed vasectomy (with azoospermia in 2 tests), 2 barrier methods (e.g., condom, diaphragm, or spermicide), or intra-uterine device];
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive;
* Able to swallow the assigned study medication tablet whole; and,
* Able to fulfill the requirements of the protocol and provide written informed consent.

Exclusion Criteria:

* History or presence of any condition or gastrointestinal (GI) surgery causing malabsorption or an effect on GI motility;
* Any uncontrolled acute disease or major surgical operation requiring hospitalization within 1 month of screening;
* History of diabetes, syncope, cardiovascular, hepatic, or renal disease;
* Uncontrolled chronic diseases such as hypertension, systemic lupus erythematosus, or rheumatoid arthritis;
* History of cancer within the last 5 years (except for basal cell carcinoma with a documented 6-month remission);
* Any known enzyme-inducer, enzyme-inhibitor, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides within 30 days of treatment;
* Any prescription drug or herbal remedy within 14 days prior to scheduled dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints of primary interest include AUC24 and the amount of 5-ASA excreted in the urine by subjects dosed with Asacol and Lialda. | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (1):
- Research Site, Miami, Florida, United States

REFERENCES:
- [Derived] Vande Casteele N, Jakate A, McNamee B, Sandborn WJ. Similar pharmacokinetics of three dosing regimens comprising two oral delayed-release mesalamine formulations in healthy adult volunteers: Randomised, open-label, parallel-group study. Br J Clin Pharmacol. 2021 Mar;87(3):1141-1149. doi: 10.1111/bcp.14479. Epub 2020 Aug 10. PMID 32671846